CLINICAL TRIAL: NCT05001932
Title: Optimizing Refractive Results and Patient Satisfaction After Cataract Surgery
Acronym: ORAPSCA
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Rigshospitalet, Denmark (Other)
Responsible Party: Principal Investigator, Anne Guldhammer Skov, MD, Medical doctor, Rigshospitalet, Denmark
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Health Services Research
Other Study IDs: H 18058722
Record Dates: First submitted 2021-08-03; First posted 2021-08-12 (Actual); Last update posted 2021-11-01 (Actual); Status verified 2021-10

CONDITIONS: Cataract
Keywords: Cataract; Anisometropia; Aniseikonia Tolerance Range
MeSH Terms: conditions — Cataract; Anisometropia | interventions — Cataract Extraction

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Multifocal (Active Comparator): Patients will receive a multifocal lens bilateral (Alcon Vivity).
  Interventions: Procedure: Cataract surgery
- Mono-vision (Active Comparator): Patients will receive a monofocal lens bilateral. Target refraction for the dominant eye will be -0.25D and for the non-dominant myopia of -2.50D.
  Interventions: Procedure: Cataract surgery
- Minimono-vision (Active Comparator): Patients will receive a monofocal lens bilateral. Target refraction for the dominant eye will be -0.25D and for the non-dominant -1.25D.
  Interventions: Procedure: Cataract surgery
- Monofocal (Active Comparator): Patients will receive a monofocal lens bilateral. Target refraction will be -0.25D.
  Interventions: Procedure: Cataract surgery

INTERVENTIONS:
Procedure: Cataract surgery — Randomized Clinical Trial

SUMMARY:
Cataract surgery is the most common eye surgery in the world. If the patient with cataract uses spectacles and both patient and surgeon find it beneficial, it is possible to compensate for the spectacles during surgery and thereby obtain a spectacle-free distance vision or spectacle-free near vision. Becoming spectacle free increases quality of life substantially and is one of the primary wishes in cataract patients. Socioeconomically, spectacle free life is beneficial as it reduces fall tendency in the elderly population. Multifocal lenses warrant the possibility of obtaining a spectacle free vision at near, intermediate and distance. It is also possible to obtain spectacle free distance and near vision or distance and intermediate vision by using traditional artificial monofocal lenses but making one eye spectacle free for distance and the other eye spectacle free for near or intermediate vision. Currently, it is not know which procedure is most beneficial for cataract patients.

In a recent PhD, the investigators developed a method, Aniseikonia Tolerance Range (ATR), that can assess how much refractive change a patient can endure without impairing stereopsis. The results demonstrated large variation in the tolerance of image difference. This method can be a future tool to assess whether a patient can tolerate the refraction that is considered most beneficial to the patient. The knowledge is important as it can help avoid improper lens choice in cataract surgery and thereby avoid stereopsis problems.

DETAILED DESCRIPTION:
Background This randomized clinical trial aims to improve visual outcomes in cataract surgery by examining which intraocular lenses (IOL)/operation methods that provide highest patient satisfaction, visual function and spectacle free vision. Furthermore, the tolerance of surgical induced refractive difference (anisometropia) will be examined and a screening method to assess how much anisometropia a patient can endure will be validated. The investigators will examine if the tolerance of anisometropia > 3 diopters is better than previously described and examine if ATR can predict which patients will experience binocular problems if exposed to surgical induced aniseikonia.These results will lead to higher patient satisfaction, better visual outcomes with elimination of patients with mediocre refractive results and visual problems due to anisometropia.

In addition the investigators will examine whether ATR is reproducible by examining the variation in the multiple measurements and in a prospective study the investigators will investigate the inter and intra person reproducibility of ATR.

100 refractive patients with healthy eyes except myopia > 3 diopters and < 6 diopters, who will have a Small Incision Lenticule Extraction (SMILE) surgery will have all investigations done. The patients will have a bilateral SMILE with a interval of seven weeks and will in between the two procedures have a surgically introduced anisometropia that will provide further knowledge on anisometropia and ATR.

ELIGIBILITY:
Inclusion Criteria:

* Bilateral cataract
* Axial length: 20-27 mm
* ACD > 2.3 mm
* Pupil size: ≥ 5.0 mm in dilatation
* Pupil siza: ≥ 2.5 mm in photo topic condition
* Stereoacuity ≤ 480 seconds of arch

Exclusion Criteria:

* Former intraocular surgery
* Other eye disease (amblyopia, strabismus, corneal pathology, glaucoma, uveitis, age related maculopathy
* Other retinal diseases
* Risk of weak zonules due to PEX or former trauma
* Astigmatism ≥ 1.0 diopter
* Diabetes
* Axial length difference between the two eyes > 0.3 mm
* Dementia
* Lack of cooperation kooperation
* Stereoacuity > 480 seconds of arc
* Complicated cataract surgery or postoperative complications (intraocular infection, retinal detachment, macular edema
* Business driving
* Night driving

Ages: 60 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 400 (Estimated)
Dates: Start 2021-08-11 (Actual); Primary Completion 2023-08-04 (Estimated); Study Completion 2024-06-01 (Estimated)

PRIMARY OUTCOMES:
Patient satisfaction | 120 days
  Investigate if MIOLs, mono-vision and mini-vision provides better visual function, quality of vision and spectacle free vision compared to monofocal IOLs. This will be evaluated by questionnaires and objective measurements as described.

SECONDARY OUTCOMES:
Tolerance of anisometropia | 120 days
  Investigate if the tolerance of anisometropia is better in the elderly population compared to a younger population (SMILE patients). This will be evaluated by questionnaires and objective measurements as described.
Aniseikonia tolerance range (ATR) | 120 days
  Compare ATR in all four arms and in a SMILE population to investigate if ATR is a future screening tool that can predict which patients cannot tolerate anisometropia
Aniseikonia tolerance range (ATR) | 120 days
  Investigate if ATR is reproducible and clinical useful in cataract patients with poor vision
Anisometropia | 120 days
  Investigate if anisometropia > 3 diopters are better tolerated than previously described. This will be evaluated by questionnaires and objective measurements as described.

CONTACTS AND LOCATIONS:
Overall Officials: Morten la Cour, MD, prof., Study Director — Glostrup University Hospital, Copenhagen
Locations (1):
- Rigshospitalet - Glostrup, Copenhagen, Glostrup, Denmark

IPD SHARING:
Plan to Share IPD: No